CLINICAL TRIAL: NCT03017560
Title: Treating Verbal Memory Deficits Following Chemotherapy for Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Shirley Ryan AbilityLab (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STU00200767
Record Dates: First submitted 2017-01-03; First posted 2017-01-11 (Estimated); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Breast Cancer Treatment; Cognitive Deficits
Keywords: Breast Cancer; Chemotherapy; Verbal Memory; Processing Speed
MeSH Terms: conditions — Cognition Disorders; Breast Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Computerized cognitive treatment (Experimental): Chosen exercises from the rehabilitation package of a commercially available, computerized, cognitive training program called Happy Neuron Pro will be used. This program was designed by a team of neurologists, neuropsychologists and cognitive psychologists, and has been successfully adapted for varying conditions of cognitive dysfunction.
  Interventions: Behavioral: Computerized cognitive treatment
- Wait list control (No Intervention): Participants assigned to the wait list control arm will receive no treatment while the experimental arm is participating in the computerized treatment. However, the computerized treatment program will be made available for these participants to utilize at the end of the study period.

INTERVENTIONS:
Behavioral: Computerized cognitive treatment — Participants will engage in auditory and verbal memory exercises intended to improve verbal memory functioning. The exercises are: Elephant Memory, Words where are you?, Split words, Bird Songs, Sound check, and You've got voicemail. Participants will complete the exercises 1 hour per day, 6 days per week, for 6 weeks. The program automatically adjusts difficulty level according to individual performance. The program captures and reports all relevant data to the primary investigator, including accuracy and reaction time (speed), which will be used to measure progress.
  Arms: Computerized cognitive treatment

SUMMARY:
The primary purpose of this study is to test the effects of a targeted, computerized cognitive training program on verbal memory in older women who have undergone chemotherapy treatment for early-stage breast cancer. As measured by neuropsychological assessment, this treatment will result in improved verbal memory. Secondarily, processing speed and naming abilities are expected to improve. Enhanced self-perception of cognitive ability is also expected.

ELIGIBILITY:
Inclusion Criteria:

* Women ages 65-90
* Chemotherapy treatment for early-stage (I, IIa, IIb, IIIa) breast cancer
* Post-menopausal
* High school education or greater
* Geographically available for followup assessment
* Native English speaker
* Normal or corrected to near-normal hearing and vision

Exclusion Criteria:

* Psychiatric history including past or current psychotic spectrum disorders (schizophrenia, bipolar disorder, major depressive disorder, dementia, schizoaffective disorder)
* Brain injury (e.g., stroke, heart attack, aneurysm, tumor, concussion, head trauma)
* Brain disease
* History of brain irradiation or surgery
* Current or past disease/disorder of the central nervous system or medical condition affecting cognitive functioning (e.g., chronic migraine, epilepsy or history of seizures, encephalitis, meningitis, multiple sclerosis, thyroid condition, Parkinson's, Alzheimer's, Huntington's disease)
* Active diagnosis of autoimmune or inflammatory disorder (e.g., systemic lupus erythematosus, rheumatoid arthritis, vasculitis, insulin-dependent diabetes, Crohn's disease, uncontrolled allergic reaction or asthma)
* History of other cancer, except for basal cell carcinoma
* Development of a second primary malignancy during the study
* Drug or alcohol abuse (i.e., more than 7 drinks per week)
* Chronic use of oral steroid medication
* Former (prior to early-stage breast cancer) intrathecal therapy, radiation therapy, chemotherapy, or any neoadjuvant chemotherapy
* Acquired or developmental speech, language, or learning disorders (e.g., aphasia, dyslexia, dysgraphia, auditory processing disorder, autism, developmental delay)
* Hormone replacement therapy, excluding vaginal estrogen

Ages: 65 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 45 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Verbal Memory | Change in Verbal Memory scores from Pretreatment/Baseline to Posttreatment/6 weeks, from Posttreatment/6 weeks to 1 month followup/10 weeks, and from Pretreatment/Baseline to 1 month followup/10 weeks.
  Immediate and delayed verbal memory

SECONDARY OUTCOMES:
Processing Speed measured via Lexical Decision Task | Change in Processing Speed scores from Pretreatment/Baseline to Posttreatment/6 weeks, from Posttreatment/6 weeks to 1 month followup/10 weeks, and from Pretreatment/Baseline to 1 month followup/10 weeks
  The Lexical Decision Task is a computerized task that measures processing speed by calculating reaction times to verb and non-verb stimuli. Outcome is measured by reaction time in milliseconds.
Processing Speed measured via Stroop Color-Word Test | Change in Processing Speed scores from Pretreatment/Baseline to Posttreatment/6 weeks, from Posttreatment/6 weeks to 1 month followup/10 weeks, and from Pretreatment/Baseline to 1 month followup/10 weeks
  The Stroop Color-Word task is a paper and pencil task that measures processing speed by assessing correct number of words read, correct number of color names read, and correct number of color-word interference pairs (i.e., names of colors printed in non-matching ink colors) read in 45 seconds. Outcomes are measured in raw scores and associated T-scores referenced against sex+age normative groups. The Stroop Color-Word Test scores will not be aggregated with the Lexical Decision Task scores.

OTHER OUTCOMES:
The Functional Assessment of Cancer Therapy-Cognition | Pre-treatment/Baseline, Post-treatment/6 weeks, 1 month followup/10 weeks
  Self-perception of cognitive ability
Treatment satisfaction survey | Pre-treatment/Baseline, Post-treatment/6 weeks, 1 month followup/10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Diane F Morean, PhD, Principal Investigator — Northwestern University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] American Cancer Society (2014). Cancer prevalence: How many people have cancer? Retrieved March 24, 2015 from http://www.cancer.org/cancer/cancerbasics/cancer-prevalence.
- [Background] McKoy JM, Samaras AT, Bennett CL. Providing cancer care to a graying and diverse cancer population in the 21st century: are we prepared? J Clin Oncol. 2009 Jun 10;27(17):2745-6. doi: 10.1200/JCO.2009.22.4352. Epub 2009 Apr 29. No abstract available. PMID 19403884
- [Background] Smith BD, Smith GL, Hurria A, Hortobagyi GN, Buchholz TA. Future of cancer incidence in the United States: burdens upon an aging, changing nation. J Clin Oncol. 2009 Jun 10;27(17):2758-65. doi: 10.1200/JCO.2008.20.8983. Epub 2009 Apr 29. PMID 19403886
- [Background] Von Ah D, Carpenter JS, Saykin A, Monahan P, Wu J, Yu M, Rebok G, Ball K, Schneider B, Weaver M, Tallman E, Unverzagt F. Advanced cognitive training for breast cancer survivors: a randomized controlled trial. Breast Cancer Res Treat. 2012 Oct;135(3):799-809. doi: 10.1007/s10549-012-2210-6. Epub 2012 Aug 24. PMID 22918524
- [Background] Poppelreuter M, Weis J, Bartsch HH. Effects of specific neuropsychological training programs for breast cancer patients after adjuvant chemotherapy. J Psychosoc Oncol. 2009;27(2):274-96. doi: 10.1080/07347330902776044. PMID 19337933
- [Background] Kesler S, Hadi Hosseini SM, Heckler C, Janelsins M, Palesh O, Mustian K, Morrow G. Cognitive training for improving executive function in chemotherapy-treated breast cancer survivors. Clin Breast Cancer. 2013 Aug;13(4):299-306. doi: 10.1016/j.clbc.2013.02.004. Epub 2013 May 4. PMID 23647804
- [Background] Ercoli LM, Castellon SA, Hunter AM, Kwan L, Kahn-Mills BA, Cernin PA, Leuchter AF, Ganz PA. Assessment of the feasibility of a rehabilitation intervention program for breast cancer survivors with cognitive complaints. Brain Imaging Behav. 2013 Dec;7(4):543-53. doi: 10.1007/s11682-013-9237-0. PMID 23955490
- [Background] Ferguson RJ, Ahles TA, Saykin AJ, McDonald BC, Furstenberg CT, Cole BF, Mott LA. Cognitive-behavioral management of chemotherapy-related cognitive change. Psychooncology. 2007 Aug;16(8):772-7. doi: 10.1002/pon.1133. PMID 17152119
- [Background] Ferguson RJ, McDonald BC, Rocque MA, Furstenberg CT, Horrigan S, Ahles TA, Saykin AJ. Development of CBT for chemotherapy-related cognitive change: results of a waitlist control trial. Psychooncology. 2012 Feb;21(2):176-86. doi: 10.1002/pon.1878. Epub 2010 Dec 2. PMID 22271538
- [Background] Lange M, Rigal O, Clarisse B, Giffard B, Sevin E, Barillet M, Eustache F, Joly F. Cognitive dysfunctions in elderly cancer patients: a new challenge for oncologists. Cancer Treat Rev. 2014 Jul;40(6):810-7. doi: 10.1016/j.ctrv.2014.03.003. Epub 2014 Mar 20. PMID 24713425
- [Background] Jenkins V, Shilling V, Fallowfield L, Howell A, Hutton S. Does hormone therapy for the treatment of breast cancer have a detrimental effect on memory and cognition? A pilot study. Psychooncology. 2004 Jan;13(1):61-6. doi: 10.1002/pon.709. PMID 14745746
- [Background] McKoy JM, Burhenn PS, Browner IS, Loeser KL, Tulas KM, Oden MR, Rupper RW. Assessing cognitive function and capacity in older adults with cancer. J Natl Compr Canc Netw. 2014 Jan;12(1):138-44. doi: 10.6004/jnccn.2014.0011. PMID 24453297
- [Background] Kueider AM, Parisi JM, Gross AL, Rebok GW. Computerized cognitive training with older adults: a systematic review. PLoS One. 2012;7(7):e40588. doi: 10.1371/journal.pone.0040588. Epub 2012 Jul 11. PMID 22792378
- [Background] Maseda A, Millan-Calenti JC, Lorenzo-Lopez L, Nunez-Naveira L. Efficacy of a computerized cognitive training application for older adults with and without memory impairments. Aging Clin Exp Res. 2013 Aug;25(4):411-9. doi: 10.1007/s40520-013-0070-5. Epub 2013 Jun 19. PMID 23780693
- [Background] Gunther VK, Schafer P, Holzner BJ, Kemmler GW. Long-term improvements in cognitive performance through computer-assisted cognitive training: a pilot study in a residential home for older people. Aging Ment Health. 2003 May;7(3):200-6. doi: 10.1080/1360786031000101175. PMID 12775401
- [Background] Smith, A. (2014). Older adults and technology use. Pew Research Center. Retrieved on March 24, 2015 from http://www.pewinternet.org/2014/04/03/older-adults-and-technology-use/.